CLINICAL TRIAL: NCT06831812
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Immunogenicity of AV-1959R in Healthy Participants
Brief Title: Phase I Clinical Study of AV-1959R: Abeta-targeting Anti-Alzheimer's Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuravax, Inc. (Industry)
Collaborators: Arvax (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AU-AV1959R-101
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Alzheimer Disease (AD); Alzheimers Disease Prevention
Keywords: vaccine; AD; prevention; precinical AD; asymptomatic AD; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm 1: AV-1959R (100 µg) + Adjuvant - Cohort 1 (Experimental): Participants receive 100 µg of AV-1959R with the adjuvant via intramuscular injection
  Interventions: Biological: AV-1959R (Abeta vaccine)
- Arm 2: Placebo (Adjuvant Only) - Cohort 1 (Experimental): Participants receive a placebo (formulation without AV-1959R) but with the adjuvant via intramuscular injection
  Interventions: Biological: AV-1959R (Abeta vaccine)
- Arm 3: AV-1959R (300 µg) + Adjuvant - Cohort 2 (Experimental): Participants receive 300 µg of AV-1959R with the adjuvant via intramuscular injection
  Interventions: Biological: AV-1959R (Abeta vaccine)
- Arm 4: Placebo (Adjuvant Only) - Cohort 2 (Experimental): Participants receive a placebo (formulation without AV-1959R) but with the adjuvant via intramuscular injection
  Interventions: Biological: AV-1959R (Abeta vaccine)

INTERVENTIONS:
Biological: AV-1959R (Abeta vaccine) — AV-1959R is an investigational adjuvanted vaccine designed to induce a targeted immune response against beta-amyloid (Aβ) to support the primary prevention of Alzheimer's disease and the treatment of asymptomatic preclinical Alzheimer's disease. It is administered intramuscularly (IM) at doses of 100 µg or 300 µg on Weeks 0, 4, and 14, in combination with the adjuvant.
  Other Names: Beta-amyloid vaccine; Aβ vaccine

SUMMARY:
This Phase 1 clinical trial evaluates the safety, tolerability, and immune response of the adjuvanted AV-1959R vaccine in healthy adults aged 40-60. Participants will receive three intramuscular injections of either adjuvanted AV-1959R (100 µg or 300 µg) or adjuvanted placebo at Weeks 0, 4, and 14, followed by an 8-week follow-up. Researchers will monitor for side effects and measure anti-Aβ antibody levels to assess immune response. This study will help determine if AV-1959R is safe and effective in generating a targeted immune response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults, 40-60 years old.
* BMI 18.0-32.0 kg/m².
* No significant medical conditions or abnormal MRI, ECG, or lab tests.
* Signed informed consent and ability to follow study procedures.
* Females must be postmenopausal or surgically sterile.
* Males must use contraception or be vasectomized.

Exclusion Criteria:

* History of Alzheimer's, stroke, or neurodegenerative disease.
* MRI abnormalities, such as infarcts or microbleeds.
* Serious illness, surgery, or hospitalization in the last 4 weeks.
* Significant heart, lung, liver, kidney, or immune disorders.
* Recent drug/alcohol abuse or severe allergies.
* Abnormal lab tests (e.g., high liver enzymes, kidney dysfunction, HIV, Hepatitis B/C positive).
* Use of investigational drugs or amyloid/tau therapies in the last year.
* Chronic use of immunosuppressants, anticoagulants, or blood products.
* Pregnant, breastfeeding, or women of childbearing potential.
* Recent blood donation (>400 mL) in the last 30 days.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of AV-1959R compared to placebo | Up to 26 weeks
  Safety and tolerability will be assessed by the incidence and severity of adverse events (AEs), serious adverse events (SAEs), and injection site reactions following intramuscular administration of AV-1959R at 100 µg and 300 µg doses.
  Safety will also be evaluated through clinical laboratory tests, vital signs, physical examinations, and MRI scans at predefined time points.

SECONDARY OUTCOMES:
Immunogenicity of AV-1959R: Anti-Aβ antibody response | Up to 26 weeks
  Immunogenicity will be assessed by quantifying anti-Aβ antibody levels in plasma samples collected at predefined study visits. Antibody titers will be determined using a validated ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Kniazev, Study Chair — Nuravax, Inc.; Hovhannes Madoyan, MD, Study Director — Arvax
Locations (1):
- Arvax, Adelaide, Australia